CLINICAL TRIAL: NCT05873621
Title: Indocyanine Green-guided Lymphadenectomy in Laparoscopic Total Mesorectal Excision for Low Rectal Cancer After Neoadjuvant Chemoradiotherapy
Acronym: (GreenEye-CRC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 279/20
Record Dates: First submitted 2023-05-04; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer; Lymph Node Cancer Metastatic
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICG-guided lymphadenectomy (Experimental): Patients will intraoperatively receive a transanal local administration of ICG. During laparoscopic total mesorectal excision, ICG-fluorescent lymph nodes beyond the mesorectum will be separately excised and sent for pathology
  Interventions: Procedure: ICG-guided lymphadenectomy

INTERVENTIONS:
Procedure: ICG-guided lymphadenectomy — Excision of ICG-fluorescent lymph nodes in addition to standard laparoscopic total mesorectal excision in rectal cancer patients after neoadjuvant chemoradiation

SUMMARY:
The goal of this clinical trial is to assess the number of harvested locoregional lymph nodes in rectal cancer patients undergoing laparoscopic total mesorectal excision and indocyanine green (ICG)-guided lymphoadenectomy after neoadjuvant chemoradiation. The main questions it aims to answer are:

* Does the use of ICG increase the total number of harvested lymph nodes?
* Does the use of ICG increase the number of harvested extra-mesorectal lymph nodes?

Participants will intraoperatively receive a trans-anal administration of ICG near to rectal cancer; during laparoscopic surgery, ICG-fluorescent nodes beyond the mesorectum will be separately excised and sent for pathology. A comparison will be performed with a recent cohort of patients affected by rectal cancer treated with standard surgery without the use of ICG.

ELIGIBILITY:
Inclusion Criteria:

* Low or middle rectal adenocarcinoma
* Indication for sphincter-saving surgery
* Neoadjuvant chemoradiation
* Indication for laparoscopic surgery
* Signed informed consent

Exclusion Criteria:

* Distant metastases at diagnosis, included peritoneal carcinomatosis
* Squamous cell cancer
* Allergy to indocyanine green

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Total number of harvested lymph nodes | 15 days
Number of harvested extra-mesorectal lymph nodes | 15 days

SECONDARY OUTCOMES:
Intraoperative and postoperative complications rates | 15 days
Time of surgery | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Cosimelli, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colletti G, Battaglia L, Sorrentino L, Guaglio M, Cosimelli M. Indocyanine green-guided lymphadenectomy of the inferior mesenteric artery in laparoscopic total mesorectal excision for low rectal cancer after neoadjuvant chemoradiotherapy - A Video Vignette. Colorectal Dis. 2022 Apr;24(4):547. doi: 10.1111/codi.16031. Epub 2022 Jan 6. No abstract available. PMID 34953173

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT05873621/Prot_SAP_000.pdf